CLINICAL TRIAL: NCT02810015
Title: Treatment of Temporo-Myofascial Disorder of Muscular Origin Using Botulinum Toxin: A Prospective Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2016:027
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Temporo-Myofascial Disorder
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botulinum Toxin A (Experimental): BTX-A will be reconstituted as directed by the manufacturer. 2.5 mL of diluent (0.9% Saline) per 100 U vial will be used to reconstitute the solution while swirling. This creates a solution with a concentration of 4 U/0.1 mL. Patients will be seated and all usual precautions of sterility and skin preparation will be completed (i.e. alcohol wipes) Injections will be administered unilateral and/or bilaterally in accordance with the topography of the corresponding muscles (temporalis and masseter) into areas of maximal tenderness and pain. Plastic single use insulin syringes with 30 gauge needles will be used to inject 30 U intramuscularly into each masseter, divided evenly into 5 sites and 20 U will be injected into each temporalis, divided evenly over 5 sites. Injections will be completed by the principal investigator and supervisors who will be trained in botulinum toxin injections.
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — BTX-A will be reconstituted as directed by the manufacturer. 2.5 mL of diluent (0.9% Saline) per 100 U vial will be used to reconstitute the solution while swirling. This creates a solution with a concentration of 4 U/0.1 mL. Patients will be seated and all usual precautions of sterility and skin preparation will be completed (i.e. alcohol wipes) Injections will be administered unilateral and/or bilaterally in accordance with the topography of the corresponding muscles (temporalis and masseter) into areas of maximal tenderness and pain. Plastic single use insulin syringes with 30 gauge needles will be used to inject 30 U intramuscularly into each masseter, divided evenly into 5 sites and 20 U will be injected into each temporalis, divided evenly over 5 sites. Injections will be completed by the principal investigator and supervisors who will be trained in botulinum toxin injections.

SUMMARY:
Temporomandibular disorders (TMD) are a group of conditions involving the temporomandibular joint (TMJ), masticatory muscles and associated structures. This broad complex of functional disorders often affects the face and jaws causing chronic pain, earaches, headaches, migraines, neck pain, and dysfunction in many people. Patients that do not find benefit with conservative management require surgical intervention. Recently, the use of botulinum toxin has proven effective and has the potential to bridge the gap between conservative therapy and surgical management resulting in less patients requiring invasive surgery. Objective: We aim to treat TMD of muscular origin using Botulinum toxin injections in the trigger points. Methods: Patients, whose pain originates from trigger points, will be enrolled in this prospective trial. This study will evaluate subjective and objective responses to treatment with botulinum toxin. The pair of masticatory muscles, masseter and temporalis, will be injected with 30 units and 20 units of botulinum toxin, respectively. Subjective outcomes such as pain and orofacial function on a visual analog scale as well as objective outcomes such as maximal interincisal mouth opening, tenderness to palpation to the temporalis and masseter muscles, maximal bite force measured by electromyogram and the reduction in muscle bulk due to muscle disuse atrophy will be assessed. Expected Results: We expect trigger points in these patients to disappear and the associated muscles to become partially paralyzed and relaxed. Consequently, we expect that the TMJ loading will be reduced and that the patient's overall functional ability will increase. We also expect that muscular hypertrophy volume from hyperactivity will decrease due to disuse atrophy and impact their cosmetic image positively. Overall, we hope these changes will result in a reduction in pain and headaches which will consequently improve the participant's diet, nutrition, psychological well being and quality of life.

DETAILED DESCRIPTION:
Introduction Temporomandibular disorders (TMD) are a group of conditions involving the temporomandibular joint (TMJ), masticatory muscles and associated structures. This broad complex of functional disorders often affects the face and jaws causing chronic pain, earaches, headaches, migraines, neck pain, and dysfunction in many people 1,2,3,4,5,6. Conservative treatment for TMD is similar to that of other musculoskeletal conditions. Pharmacologic therapy includes the use of anti-inflammatory medications, muscle relaxants, or opioid analgesics7,8,9,10. Physical treatments comprise of dental splints, directed physiotherapy, moist heat therapy, soft diet, massage and acupuncture11,12,13,14,15,16,17,18,19,20,21,22,23,24,25. At the extreme end of the spectrum, surgical management includes arthrocentesis, arthroscopy and open joint procedures26,27,28,29,30,31,32,33,34,35,36,37,38,39,40,41,42,43,44. Some patients can find relief with a combination of these previously mentioned interventions; however, none of these have been proven to be consistently effective. Open joint procedures are not reversible while anti-inflammatory medications and narcotics can have undesirable side effects on the gastrointestinal and central nervous system, respectively. Furthermore, many patients suffering from severe chronic pain do not feel relief with even the strongest narcotic analgesics45,46.

TMD has a complex etiology consisting of components from internal derangement of the joint, arthralgia and/or a component of myofascial pain and muscle hyperactivity1,2,3,4. A treatment that has high specificity and low side effects directed solely at the muscular aspect, which presents with signs and symptoms of trigger points, clenching, and bruxism, could produce another avenue of intervention with significant potential. Recently, the use of botulinum toxin has proven effective and has the potential to be such an agent for treatment with patients suffering from TMD and other orofacial pain conditions47,48,49,50,51,52,53,54,55.

Botulinum toxins are exotoxins derived from Clostridium botulinum, a gram-positive, anaerobic, spore-forming organism. There are 8 different subtypes; type A (BTX-A) has been used in recent studies for the treatment of motor disorders such as cervical dystonia or the hyperactive muscular component of TMD53,54,55. The specific method of action of botulinum toxin is on peripheral synapses. In the synaptic cleft, the botulinum toxin is brought into the presynaptic cell by endocytosis. It acts by blocking the calcium induced release of acetylcholine by selective proteolysis of synaptomal-associated proteins (SNAP)47,48,4,50,51,52,53,54,55. Inhibition of acytelcholine thus causes an inhibition of muscular hyperactivity.

Botulinum toxin has a number of indications approved by the Food and Drug Administration such as the therapeutic treatment for cervical dystonia, cosmetic use such as glabellar lines and wide spectrum of off-label uses such as extracervical spasticities, cerebral palsy, post stroke spasticity, neurologic, dermatologic, and gastrointestinal disorders56. Off-label use of a licensed drug or biologic product occurs with a wide range of products57,58,59.

Objective of the Study We aim to treat TMD of muscular origin using Botulinum toxin injections in the trigger points.

Method Our study will enroll selective patients attending the Oral and Maxillofacial Surgery clinic at the Health Sciences Center and at the University of Manitoba College of Dentistry over a 2-year period. Subjects will be recruited from referrals coming to the Health Sciences Center and College of Dentistry. The design will be prospective study following subjective outcomes such as pain and orofacial function on a visual analog scale as well as objective outcomes such as maximal interincisal mouth opening, tenderness to palpation to the temporalis and masseter muscles, maximal bite force measured by electromyogram and the reduction in muscle bulk due to muscle disuse atrophy. These outcomes have an appreciable affect on the patient's quality of life and provide subjective and objective measurements for analysis and study.

Inclusion criteria for patient's enrolled in this study include: participant's with trigger points in their masticatory muscles including, but not limited to: masseter and temporalis either bilateral or unilateral and secondly, have tried conservative management for at least 3 months and have shown to be refractory to these interventions. Exclusion criteria include: participant's that do not satisfy the inclusion criteria, currently are breastfeeding or pregnant, participant's whose TMD is not muscular in origin, inability to speak or understand English, the inability to provide meaningful informed consent due to physical, cognitive or psychiatric disability, a previous known allergy to Botulinum toxin, multiple sclerosis, pre-existing neuromuscular disorders, Lambert-Eaton syndrome, or chronic centrally mediated neuralgic pain patients.

Before enrollment, informed consent will be obtained from each patient. Informed consent will consist of a thorough initial evaluation and interview. If the patient is assessed to be appropriate for the study the patient will be informed of all risks and potential consequences of the study. Additional information will be given regarding benefits, cost and time required. During the informed consent, the principal investigator and at least one supervisor will be in attendance to answer any questions. Patients will be allowed time to think about their decision and discuss with family members and their family physician. A future appointment can be made to obtain consent and will be witnessed by the principal investigator, a supervisor and an OMFS assistant that has no connection with the study.

On the initial assessment, multiple measurements will be taken (see clinical assessment form attached). Additionally, an appointment will be made for the patient to have their maximal bite force registered pre-injection with the use of EMG.

BTX-A will be reconstituted as directed by the manufacturer. 2.5 mL of diluent (0.9% Saline) per 100 U vial will be used to reconstitute the solution while swirling. This creates a solution with a concentration of 4 U/0.1 mL. Patients will be seated and all usual precautions of sterility and skin preparation will be completed (i.e. alcohol wipes) Injections will be administered unilateral and/or bilaterally in accordance with the topography of the corresponding muscles (temporalis and masseter) into areas of maximal tenderness and pain. Plastic single use insulin syringes with 30 gauge needles will be used to inject 30 U intramuscularly into each masseter, divided evenly into 5 sites and 20 U will be injected into each temporalis, divided evenly over 5 sites. Injections will be completed by the principal investigator and supervisors who will be trained in botulinum toxin injections.

Patients will have scheduled follow ups at 1 week, 1 month, 3 months and 6 months post-injection. An additional follow up call will be made the next day after injection. The clinical assessment form will be used by the principal investigator to take measurements at each follow up appointment, except EMG readings which will only be done at the initial assessment and 3 month follow up appointment. This will provide a total of 5 assessments (including the initial assessment). During this time period, patients will be asked to stop any treatment for their TMD other than analgesics as required.

Subjective pain scores will be assessed on a visual analog scale (VAS) where 0 is no pain and 10 is the worst facial or jaw pain they've ever experience. Subjective functional assessments will also be assessed with VAS where 0 means no limitation and 10 indicates severe limitation with scales for chewing, drinking, exercising, eating hard food, eating soft food, smiling or laughing, cleaning their teeth, yawning, swallowing and talking. Objectively, range of motion will be assessed with a Boley gauge between the same upper and lower incisor each time. Palpation tenderness will be objectively assessed in bilateral temporalis and masseter muscles. Pain to pressure will be ranked from 0 to 5, with 0 indicating no pain and 5 representing extreme debilitating pain. Addition of each score will give a composite score of the overall facial tenderness out of a maximal score of 24 (2 areas X 6 scores X bilaterally). All assessments will be completed by the same examiner every time at the same time of day. Lastly, a measurement of the facial width will be taken. A point inferior to each ear lobule bilaterally will be marked as well as a point on the menton will be chosen and recorded. The distance unilaterally from one lobule to menton will be measured for left and right sides and a total distance will also be calculated to assess facial width. This will be used to determine the cosmetic change due to disuse atrophy 60.

Side effects may include, but are not limited to: transient facial asymmetry during dynamic movements, dysphagia, ptosis, erythematous discoloration or edema at the injection site, rash, and difficulty chewing hard food 61. Every attempt will be made to insure injection of the botulinum in the appropriate site. Aspiration before each injection will help prevent any intravascular and systemic effects while proper patient positioning and proper site identification will help prevent unwanted side effects such as ptosis. If a rash develops, Benadryl will be the first line medication given immediately followed by a several day course of Benadryl at home. In the case of an emergent reaction, adequate management would be undertaken at the clinic and referral to an appropriate service if necessary. Due to passage across the placenta, the use during pregnancy is also contraindicated. All patient's who are currently breastfeeding or pregnant will be excluded from the study62.

Funding for the study will be provided by application to research grants through The University of Manitoba and the Canadian Association of Oral and Maxillofacial Surgeons.

Anticipated results We expect trigger points in these patients to disappear and the associated muscles to become partially paralyzed and relaxed. Consequently, we expect that the TMJ loading will be reduced and that the patient's overall functional ability will increase. We also expect that muscular hypertrophy volume from hyperactivity will decrease due to disuse atrophy and impact their cosmetic image positively. Overall, we hope these changes will result in a reduction in pain and headaches which will consequently improve the participant's diet, nutrition, psychological well being and quality of life.

We expect this study will be published in the International Journal of Oral and Maxillofacial Surgery and that results will be presented at the International meeting of Oral and Maxillofacial Surgeons in 2018.

ELIGIBILITY:
Inclusion Criteria:

* Participant's with trigger points in their masticatory muscles including, but not limited to: masseter and temporalis either bilateral or unilateral and secondly
* have tried conservative management for at least 3 months and have shown to be refractory to these interventions.

Exclusion Criteria:

* participant's that do not satisfy the inclusion criteria
* currently are breastfeeding or pregnant
* participant's whose TMD is not muscular in origin
* inability to speak or understand English
* the inability to provide meaningful informed consent due to physical, cognitive or psychiatric disability
* a previous known allergy to Botulinum toxin
* multiple sclerosis
* pre-existing neuromuscular disorders
* Lambert-Eaton syndrome
* chronic centrally mediated neuralgic pain patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Pain (Visual Analog Scale) | 3 months
  Subjective pain scores will be assessed on a visual analog scale (VAS) where 0 is no pain and 10 is the worst facial or jaw pain they've ever experience. Subjective functional assessments will also be assessed with VAS where 0 means no limitation and 10 indicates severe limitation with scales for chewing, drinking, exercising, eating hard food, eating soft food, smiling or laughing, cleaning their teeth, yawning, swallowing and talking.
Range of Motion | 3 months
  Range of motion will be assessed with a Boley gauge between the same upper and lower incisor each time
Palpation tenderness | 3 months
  Pain to pressure will be ranked from 0 to 5, with 0 indicating no pain and 5 representing extreme debilitating pain. Addition of each score will give a composite score of the overall facial tenderness out of a maximal score of 24 (2 areas X 6 scores X bilaterally).

SECONDARY OUTCOMES:
Facial Width | 3 months
  A point inferior to each ear lobule bilaterally will be marked as well as a point on the menton will be chosen and recorded. The distance unilaterally from one lobule to menton will be measured for left and right sides and a total distance will also be calculated to assess facial width.

CONTACTS AND LOCATIONS:
Overall Officials: Reda Elgazzar, DMD, Study Director — University of Manitoba

REFERENCES:
- [Background] Kaplan AS, Assael LA. Temporomandibular disorders: diagnosis and treatment. Philadelphia (PA): W.B. Saunders Company; 1991. p. 522-5.
- [Background] Travell JG, Simons DG. Myofascial pain and dysfunction: the trigger point manual. Baltimore (MD):Williams & Wilkins; 1983.
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Adler RC, Adachi NY. Physical medicine in the management of myofascial pain and dysfunction: medical management of temporomandibular disorders. Oral Maxillofac Surg Clin North Am 1995;7(1):99-106.
- [Background] Gangarosa LP, Mahan PE. Pharmacologic management of TMJ-MPDS. Ear Nose Throat J 1982;61:670.
- [Background] Murphy GJ. Physical medicine modalities and trigger point injections in the management of temporomandibular disorders and assessing treatment outcome. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1997 Jan;83(1):118-22. doi: 10.1016/s1079-2104(97)90101-3. PMID 9007934
- [Background] Syrop S. Pharmacologic management of myofascial pain and dysfunction.Oral Maxillofac Surg Clin North Am 1995;7:87-97.
- [Background] Dimitroulis G, Gremillion HA, Dolwick MF, Walter JH. Temporomandibular disorders. 2. Non-surgical treatment. Aust Dent J. 1995 Dec;40(6):372-6. doi: 10.1111/j.1834-7819.1995.tb04835.x. PMID 8615742
- [Background] Yoshida H, Fukumura Y, Fujita S, Nishida M, Iizuka T. The expression of cyclooxygenase-2 in human temporomandibular joint samples: an immunohistochemical study. J Oral Rehabil. 2002 Dec;29(12):1146-52. doi: 10.1046/j.1365-2842.2002.00969.x. PMID 12472850
- [Background] Quinn JH, Kent JH, Moise A, Lukiw WJ. Cyclooxygenase-2 in synovial tissue and fluid of dysfunctional temporomandibular joints with internal derangement. J Oral Maxillofac Surg. 2000 Nov;58(11):1229-32; discussion 1232-3. doi: 10.1053/joms.2000.16619. PMID 11078133
- [Background] Israel HA, Syrop SB. The important role of motion in the rehabilitation of patients with mandibular hypomobility: a review of the literature. Cranio. 1997 Jan;15(1):74-83. doi: 10.1080/08869634.1997.11745995. PMID 9586491
- [Background] Karlis V, Andreopoulos N, Kinney L, Glickman R. Effectiveness of supervised calibrated exercise therapy on jaw mobility and temporomandibular dysfunction. J Oral Maxillofac Surg 1994;52(8 Suppl 2):147.
- [Background] Sebastian MH, Moffett BC. The effects of continuous passive motion on the temporomandibular joint after surgery. Part II. Appliance improvement, normal subject evaluation, pilot clinical trial. Oral Surg Oral Med Oral Pathol. 1989 Jun;67(6):644-53. doi: 10.1016/0030-4220(89)90002-9. PMID 2662104
- [Background] Maloney GE, Mehta N, Forgione AG, Zawawi KH, Al-Badawi EA, Driscoll SE. Effect of a passive jaw motion device on pain and range of motion in TMD patients not responding to flat plane intraoral appliances. Cranio. 2002 Jan;20(1):55-66. doi: 10.1080/08869634.2002.11746191. PMID 11831346
- [Background] Yuasa H, Kurita K; Treatment Group on Temporomandibular Disorders. Randomized clinical trial of primary treatment for temporomandibular joint disk displacement without reduction and without osseous changes: a combination of NSAIDs and mouth-opening exercise versus no treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Jun;91(6):671-5. doi: 10.1067/moe.2001.114005. PMID 11402280
- [Background] Moses JJ, Sartoris D, Glass R, Tanaka T, Poker I. The effect of arthroscopic surgical lysis and lavage of the superior joint space on TMJ disc position and mobility. J Oral Maxillofac Surg. 1989 Jul;47(7):674-8. doi: 10.1016/s0278-2391(89)80004-7. PMID 2732826
- [Background] Nelson SJ, Ash MM Jr. An evaluation of a moist heating pad for the treatment of TMJ/muscle pain dysfunction. Cranio. 1988 Oct;6(4):355-9. doi: 10.1080/08869634.1988.11678261. No abstract available. PMID 3255522
- [Background] Matsumura WM. Use of acupressure techniques and concepts for nonsurgical management of TMJ disorders. J Gen Orthod. 1993 Mar;4(1):5-16. No abstract available. PMID 8399726
- [Background] Elsharkawy TM, Ali NM. Evaluation of acupuncture and occlusal splint therapy in the treatment of temporomandibular joint disorders. Egypt Dent J. 1995 Jul;41(3):1227-32. PMID 9497660
- [Background] Berry H, Fernandes L, Bloom B, Clark RJ, Hamilton EB. Clinical study comparing acupuncture, physiotherapy, injection and oral anti-inflammatory therapy in shoulder-cuff lesions. Curr Med Res Opin. 1980;7(2):121-6. doi: 10.1185/03007998009112038. PMID 7002481
- [Background] Okeson JP, Kemper JT, Moody PM. A study of the use of occlusion splints in the treatment of acute and chronic patients with craniomandibular disorders. J Prosthet Dent. 1982 Dec;48(6):708-12. doi: 10.1016/s0022-3913(82)80034-6. PMID 6961210
- [Background] Okeson JP, Moody PM, Kemper JT, Haley JV. Evaluation of occlusal splint therapy and relaxation procedures in patients with temporomandibular disorders. J Am Dent Assoc. 1983 Sep;107(3):420-4. doi: 10.14219/jada.archive.1983.0275. PMID 6355230
- [Background] Clark GT. A critical evaluation of orthopedic interocclusal appliance therapy: design, theory, and overall effectiveness. J Am Dent Assoc. 1984 Mar;108(3):359-64. doi: 10.14219/jada.archive.1984.0010. PMID 6371096
- [Background] Rugh JD, Harlan J. Nocturnal bruxism and temporomandibular disorders. Adv Neurol. 1988;49:329-41. PMID 3278546
- [Background] Okeson JP. Occlusal appliance therapy. In: Duncan LL, editor. Management of temporomandibular disorders and occlusion. 4th ed. Philadelphia (PA): Mosby Publishing; 1998. p. 474-502.
- [Background] Major PW, Nebbe B. Use and effectiveness of splint appliance therapy: review of literature. Cranio. 1997 Apr;15(2):159-66. doi: 10.1080/08869634.1997.11746007. PMID 9586519
- [Background] Nitzan DW, Price A. The use of arthrocentesis for the treatment of osteoarthritic temporomandibular joints. J Oral Maxillofac Surg. 2001 Oct;59(10):1154-9; discussion 1160. doi: 10.1053/joms.2001.26716. PMID 11573170
- [Background] Bronstein SL, Thomas M. Arthroscopy of the temporomandibular joint. Philadelphia (PA):W.B. Saunders Co.; 1991. p. 320.
- [Background] Goss AN, Bosanquet AG. Temporomandibular joint arthroscopy. J Oral Maxillofac Surg. 1986 Aug;44(8):614-7. doi: 10.1016/s0278-2391(86)80072-6. PMID 3461140
- [Background] Sanders B, Buoncristiani R. Diagnostic and surgical arthroscopy of the temporomandibular joint: clinical experience with 137 procedures over a 2-year period. J Craniomandib Disord. 1987 Fall;1(3):202-13. No abstract available. PMID 3481380
- [Background] Holmlund A, Hellsing G. Arthroscopy of the temporomandibular joint. An autopsy study. Int J Oral Surg. 1985 Apr;14(2):169-75. doi: 10.1016/s0300-9785(85)80089-2. PMID 3920161
- [Background] Ohnishi M. Clinical application of arthroscopy in the temporomandibular joint diseases. Bull Tokyo Med Dent Univ. 1980 Sep;27(3):141-50. PMID 6936091
- [Background] Onishi M. [Arthroscopy of the temporomandibular joint (author's transl)]. Kokubyo Gakkai Zasshi. 1975 Jun;42(2):207-13. No abstract available. Japanese. PMID 1058272
- [Background] Dolwick MF, Riggs RR. Diagnosis and treatment of internal derangements of the temporomandibular joint. Dent Clin North Am. 1983 Jul;27(3):561-72. No abstract available. PMID 6578966
- [Background] McCarty WL, Farrar WB. Surgery for internal derangements of the temporomandibular joint. J Prosthet Dent. 1979 Aug;42(2):191-6. doi: 10.1016/0022-3913(79)90174-4. PMID 287798
- [Background] Moses JJ, Poker ID. TMJ arthroscopic surgery: an analysis of 237 patients. J Oral Maxillofac Surg. 1989 Aug;47(8):790-4. doi: 10.1016/s0278-2391(89)80035-7. PMID 2746386
- [Background] Moses JJ, Lo HH, Lee J, Topper DC. Tomographic changes in the temporomandibular joint following arthroscopic surgery with lysis and lavage and eminentia release. J Orofac Pain. 1994 Fall;8(4):407-12. PMID 7670430
- [Background] Walker RV, Kalamchi S. A surgical technique for management of internal derangement of the temporomandibular joint. J Oral Maxillofac Surg. 1987 Apr;45(4):299-305. doi: 10.1016/0278-2391(87)90347-8. PMID 3470447
- [Background] Hall MB. Meniscoplasty of the displaced temporomandibular joint meniscus without violating the inferior joint space. J Oral Maxillofac Surg. 1984 Dec;42(12):788-92. doi: 10.1016/0278-2391(84)90346-x. PMID 6594472
- [Background] Weinberg S. Eminectomy and meniscorhaphy for internal derangements of the temporomandibular joint. Rationale and operative technique. Oral Surg Oral Med Oral Pathol. 1984 Mar;57(3):241-9. doi: 10.1016/0030-4220(84)90177-4. PMID 6584814
- [Background] Eriksson L, Westesson PL. Diskectomy in the treatment of anterior disk displacement of the temporomandibular joint. A clinical and radiologic one-year follow-up study. J Prosthet Dent. 1986 Jan;55(1):106-16. doi: 10.1016/0022-3913(86)90085-5. No abstract available. PMID 3456042
- [Background] Kondoh T, Hamada Y, Kamei K, Seto K. Simple disc reshaping surgery for internal derangement of the temporomandibular joint: 5-year follow-up results. J Oral Maxillofac Surg. 2003 Jan;61(1):41-8; discussion 48. doi: 10.1053/joms.2003.50007. PMID 12524606
- [Background] Zenz M, Strumpf M, Tryba M. Long-term oral opioid therapy in patients with chronic nonmalignant pain. J Pain Symptom Manage. 1992 Feb;7(2):69-77. doi: 10.1016/0885-3924(92)90116-y. PMID 1573287
- [Background] Zuniga JR. The use of nonopioid drugs in management of chronic orofacial pain. J Oral Maxillofac Surg. 1998 Sep;56(9):1075-80. doi: 10.1016/s0278-2391(98)90260-9. PMID 9734770
- [Background] Tan EK, Jankovic J. Treating severe bruxism with botulinum toxin. J Am Dent Assoc. 2000 Feb;131(2):211-6. doi: 10.14219/jada.archive.2000.0149. PMID 10680389
- [Background] Freund B, Schwartz M, Symington JM. Botulinum toxin: new treatment for temporomandibular disorders. Br J Oral Maxillofac Surg. 2000 Oct;38(5):466-71. doi: 10.1054/bjom.1999.0238. PMID 11010775
- [Background] Freund B, Schwartz M. The use of botulinum toxin for the treatment of temporomandibular disorder. Oral Health. 1998 Feb;88(2):32-7. No abstract available. PMID 9610334
- [Background] Borodic GE, Acquadro MA. The use of botulinum toxin for the treatment of chronic facial pain. J Pain. 2002 Feb;3(1):21-7. doi: 10.1054/jpai.2002.27142. PMID 14622850
- [Background] Ziegler CM, Haag C, Muhling J. Treatment of recurrent temporomandibular joint dislocation with intramuscular botulinum toxin injection. Clin Oral Investig. 2003 Mar;7(1):52-5. doi: 10.1007/s00784-002-0187-y. Epub 2003 Jan 25. PMID 12673439
- [Background] Karacalar A, Yilmaz N, Bilgici A, Bas B, Akan H. Botulinum toxin for the treatment of temporomandibular joint disk disfigurement: clinical experience. J Craniofac Surg. 2005 May;16(3):476-81. doi: 10.1097/04.scs.0000157263.73768.64. PMID 15915120
- [Background] Freund BJ, Schwartz M. Relief of tension-type headache symptoms in subjects with temporomandibular disorders treated with botulinum toxin-A. Headache. 2002 Nov-Dec;42(10):1033-7. doi: 10.1046/j.1526-4610.2002.02234.x. PMID 12453036
- [Background] von Lindern JJ, Niederhagen B, Berge S, Appel T. Type A botulinum toxin in the treatment of chronic facial pain associated with masticatory hyperactivity. J Oral Maxillofac Surg. 2003 Jul;61(7):774-8. doi: 10.1016/s0278-2391(03)00153-8. PMID 12856249
- [Background] von Lindern JJ. Type A botulinum toxin in the treatment of chronic facial pain associated with temporo-mandibular dysfunction. Acta Neurol Belg. 2001 Mar;101(1):39-41. PMID 11379274
- [Background] Cote TR, Mohan AK, Polder JA, Walton MK, Braun MM. Botulinum toxin type A injections: adverse events reported to the US Food and Drug Administration in therapeutic and cosmetic cases. J Am Acad Dermatol. 2005 Sep;53(3):407-15. doi: 10.1016/j.jaad.2005.06.011. PMID 16112345
- [Background] Kocs D, Fendrick AM. Effect of off-label use of oncology drugs on pharmaceutical costs: the rituximab experience. Am J Manag Care. 2003 May;9(5):393-400; quiz 401-2. PMID 12744301
- [Background] Stone KJ, Viera AJ, Parman CL. Off-label applications for SSRIs. Am Fam Physician. 2003 Aug 1;68(3):498-504. PMID 12924832
- [Background] Off-label use of tumor necrosis factor inhibitors on ankylosing spondylitis, ulcerative colitis, and psoriasis. TEC Bull (Online). 2003 Jun 3;20(2):9-18. No abstract available. PMID 12854551
- [Background] Kim HJ, Yum KW, Lee SS, Heo MS, Seo K. Effects of botulinum toxin type A on bilateral masseteric hypertrophy evaluated with computed tomographic measurement. Dermatol Surg. 2003 May;29(5):484-9. doi: 10.1046/j.1524-4725.2003.29117.x. PMID 12752515
- [Background] Ihde SK, Konstantinovic VS. The therapeutic use of botulinum toxin in cervical and maxillofacial conditions: an evidence-based review. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Aug;104(2):e1-11. doi: 10.1016/j.tripleo.2007.02.004. Epub 2007 Jun 7. PMID 17560141
- [Background] Umstadt HE. [Botulinum toxin in oromaxillofacial surgery]. Mund Kiefer Gesichtschir. 2002 Jul;6(4):249-60. doi: 10.1007/s10006-002-0390-7. German. PMID 12242934